CLINICAL TRIAL: NCT02459756
Title: Effects of an Anthocyanin-rich Blackcurrant Beverage on Cardiovascular Function
Brief Title: Anthocyanin-rich Blackcurrant and Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Professor Parveen Yaqoob, MA, DPhil, RNutr, FAfN, Professor Parveen Yaqoob, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: UREC 14/17
Record Dates: First submitted 2015-05-20; First posted 2015-06-02 (Estimated); Last update posted 2016-02-09 (Estimated); Status verified 2016-02

CONDITIONS: Vascular Stiffness; Inflammation
Keywords: anthocyanins; bioavailability
MeSH Terms: conditions — Inflammation | interventions — Water; Sucrose; Glucose; Fructose; maltodextrin; malic acid; Citric Acid; Ascorbic Acid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Active Comparator): Spray dried blackcurrant powder dissolved in water
  Interventions: Other: Beverage: Spray dried blackcurrant powder dissolved in water
- Placebo (Placebo Comparator): (sucrose, glucose, fructose, maltodextrin, malic acid, citric acid, vitamin C, artificial blackcurrant flavouring and low-nitrate water)
  Interventions: Other: Beverage: Placebo (sucrose, glucose, fructose, maltodextrin, malic acid, citric acid, vitamin C, artificial blackcurrant flavouring and low-nitrate water)

INTERVENTIONS:
Other: Beverage: Spray dried blackcurrant powder dissolved in water
  Arms: Intervention
Other: Beverage: Placebo (sucrose, glucose, fructose, maltodextrin, malic acid, citric acid, vitamin C, artificial blackcurrant flavouring and low-nitrate water)
  Arms: Placebo

SUMMARY:
Regular consumption of fruits and vegetables may improve human health and reduce the risk of chronic diseases, such as heart disease, certain cancers and type 2 diabetes, but the active components and the underlying mechanisms are poorly understood. Berry fruits are abundant in anthocyanins and this study aims to test the hypothesis that ingestion of an anthocyanin-rich blackcurrant beverage will improve markers of cardiovascular health (health of blood vessels, inflammation and platelet function). Further, the study will investigate the anthocyanin bioavailability from the blackcurrant beverage.

ELIGIBILITY:
Inclusion Criteria:

* Aged 30-55 years
* Non-smoker
* BMI between 20 - 30 kg/m2
* Generally healthy as established by a 'health and lifestyle' questionnaire and a screening blood sample
* Blood pressure < 140/90mmHg
* Total cholesterol < 6.2 mmol/L
* Fasting glucose < 7.0 mmol/L

Exclusion Criteria:

* Diabetes mellitus
* Heart problems, stroke, vascular disease
* Inflammatory disease
* Kidney, liver, pancreas or gastrointestinal diseases
* Medication for hyperlipidaemia, hypertension, hypercoagulation, inflammatory conditions
* Asthma
* Allergies
* Smokers (social smokers who agree to abstain for 1 month before and during the study not excluded)
* Taking phytochemical, antioxidant or fish oil supplements (unless willing to stop for the study period)
* Taking aspirin > 2 times per month and unwilling to abstain from aspirin ingestion for 14 days prior each study visit
* History of alcohol misuse
* Consumption of alcohol >21 units (men) or >15 units (women)
* Vegans
* Intense aerobic exercise >20 min 3 x per week
* Participation in another clinical trial
* Antibiotics in previous 3 months before study
* Low haemoglobin levels
* Females who are pregnant, lactating, or if of reproductive age and not using a reliable form of contraception (including abstinence)

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2015-06; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in vascular reactivity measured by flow-mediated dilatation (FMD) | Acute study: measured at baseline and 1, 2, 4 and 6 h post intervention
Change from baseline in platelet function measured by agonist-induced platelet aggregation | Acute study: measured at baseline and 2 and 4 h post intervention

SECONDARY OUTCOMES:
Change from baseline in the concentration of polyphenols and their metabolites and degradants in blood and urine samples measured by HPLC-MS/MS | Acute study: plasma measured at baseline and 1, 2, 4, 6 and 24 h post intervention, urine measured at baseline and 1, 2, 4, 6 and 6-24 h post intervention
Change from baseline in vascular function measured by digital volume pulse (DVP) | Acute study: measured at baseline and 2, 4 and 6 h post intervention
Change from baseline in blood pressure | Acute study: measured at baseline and 1, 2, 4 and 6 h post intervention
Change from baseline in the concentration of nitric oxide in plasma measured by ozone-based chemiluminescence | Acute study: measured at baseline and 1, 2, 4 and 6 h post intervention
Change from baseline in the concentration of selected cytokines (TNF-a, IL-1b, IL-6, IL-8 and IL-10) in plasma measured using a cytometric bead array kit from BD Biosciences | Acute study: measured at baseline and 1, 2, 4 and 6 h post intervention
Change from baseline in platelet function (numbers of circulating micro particles by nano particle tracking analysis) | Acute study: measured at baseline and 1, 2, 4 and 6 h post intervention (urine metabonomics additionally 6-24h)
Metabonomics on urine and plasma samples measured by nuclear magnetic resonance spectroscopy | Acute study: measured at baseline and 1, 2, 4 and 6 h post intervention (urine metabonomics additionally 6-24h)

CONTACTS AND LOCATIONS:
Overall Officials: Parveen Yaqoob, DPhil, Principal Investigator — University of Reading
Locations (1):
- University of Reading, Reading, United Kingdom

REFERENCES:
- [Derived] Amini AM, Zhou R, Austermann K, Kralova D, Serra G, Ibrahim IS, Corona G, Bergillos-Meca T, Aboufarrag H, Kroon PA, Spencer JP, Yaqoob P. Acute Effects of an Anthocyanin-Rich Blackcurrant Beverage on Markers of Cardiovascular Disease Risk in Healthy Adults: A Randomized, Double-Blind, Placebo-Controlled, Crossover Trial. J Nutr. 2025 Jul;155(7):2275-2289. doi: 10.1016/j.tjnut.2025.05.017. Epub 2025 May 23. PMID 40414296